CLINICAL TRIAL: NCT04221685
Title: Intraoperative Pain During Extraction of Maxillary Primary Molars Using Artpharma Versus Artinibsa in Children After Infiltration Technique: a Randomized Clinical Trial
Brief Title: Intraoperative Pain After Infiltration Technique Using Artpharma Versus Artinibsa in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hafedha Hashem Abdullah, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IOP Use Artp Vs Artin inf
Record Dates: First submitted 2020-01-01; First posted 2020-01-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pain, Postoperative
Keywords: Articaine; Extraction primary teeth; Infiltration technique; Postoperative pain; Intraoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant) single ( participant ) because the two interventions used in this trial are easily recognized by the investigator but the participant and the statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artinibsa (Active Comparator): Powerful local anaesthetic with a short latency time. Its high lipid solubility gives it better diffusion through soft tissues and bone and makes it highly effective for infiltrative techniques.4%Articaine 1:100000.
  Interventions: Other: Artinibsa
- Artpharma (Experimental): ArtPharma is a unique amide local anesthetic that is currently Used in dentistry Amides has taken over their predecessors esters with their enhanced performance.Each ml Articaine (D.C.I) 40.00 mg hydrochloride,Epinephrine (D.C.I) (tartrate) 0.01 mg
  Interventions: Other: Artpharma

INTERVENTIONS:
Other: Artpharma — ArtPharma is a unique amide local anesthetic that is currently Used in dentistry Amides has taken over their predecessors esters with their enhanced performance.Each ml Articaine (D.C.I) 40.00 mg hydrochloride, Epinephrine (D.C.I) (tartrate) 0.01 mg
  Arms: Artpharma
Other: Artinibsa — Powerful local anaesthetic with a short latency time.
  Its high lipid solubility gives it better diffusion through soft tissues and bone and makes it highly effective for infiltrative techniques.Each ml contains:
  Articaine (D.C.I) 40.00 mg hydrochloride, Epinephrine (D.C.I) (tartrate) 0.01 mg
  Arms: Artinibsa

SUMMARY:
The aim of this study is to assess Intraoperative pain for extraction of Maxillary primary molars using Artpharma Versus Artinibsa in children during infiltration technique.

DETAILED DESCRIPTION:
Articaine is used for pain control Like other local anesthetic drugs, articaine causes a temporary and completely reversible state of anesthesia (loss of sensation) during (dental) procedures.This local anesthesia was first synthesized by Rusching in 1969, and carried to the market in Germany by Hoechst AG, a life-sciences German company, under the brand name Ultracain ,it entered clinical practice in Germany in 1976. The name was changed in 1984, the year it was released in Canada. It then entered the United Kingdom in 1998, the United States in 2000 and Australia in 2005. At this time, articaine is available as a 4% solution containing 1:100, 000 or 1:200, 000 adrenaline. Articaine has been widely used in dental surgery.It started to use carticaine around 1977.In dentistry has been investigated widely. Articaine is a unique amide LA in that it contains a thiophene, instead of a benzene ring.The thiophene ring allows greater lipid solubility and effectiveness as a greater portion of an administered dose can enter neurons

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-9 years.
* Children with maxillary primary molars indicated for extraction.

Exclusion Criteria:

* Children with medical conditions.
* Uncooperative children.
* Parents or guardians who refuse participating in the study.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — 6-9years
Enrollment: 130 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative pain. | immediate
  Intraoperative pain: is measuring by using Wong Baker visual analogue scale and measuring unite is Scale (0-10).

SECONDARY OUTCOMES:
Pain during injection(success rate). | immediate
  Pain during injection:is evaluated the success rate of anesthesia by using the visual analogue scale and measuring unite is categorical.
Onset of anesthesia. | Immediate
  onset of anesthesia:is measuring by using stop watch and the unit is minutes
The sensation after injection. | Immediate
  The sensation after injection: is evaluated the effect of the anesthesia by checking mucous using the probe and measuring unite is binary (Yes or No).

IPD SHARING:
Plan to Share IPD: No